CLINICAL TRIAL: NCT04355598
Title: Comparative Safety and Efficacy of Cervical Lidocaine-Prilocaine Cream Versus Glyceryl Trinitrate Cream on Pain Perception During Levonorgestrel- Intrauterine Device Insertion Among Nulliparous Women: a Randomized Double-blind Controlled Trial
Brief Title: Cervical Lidocaine-Prilocaine Cream vs Glyceryl Trinitrate Cream in Nulliparous Women With LNG-IUD Insertion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: glyceryl trinitrate IUD
Record Dates: First submitted 2020-04-18; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine-Prilocaine cream (Experimental): 2 mL of the Lidocaine-Prilocaine cream will be placed on the anterior lip of the cervix by a Q-tip applicator, followed by 2 mL will be introduced in the cervical canal 7 minutes prior to IUD insertion
  Interventions: Drug: Lidocaine-Prilocaine cream
- glyceryl trinitrate cream (Active Comparator): 2 mL of the glyceryl trinitrate cream will be placed on the anterior lip of the cervix by a Q-tip applicator, followed by 2 mL will be introduced in the cervical canal 7 minutes prior to IUD insertion
  Interventions: Drug: glyceryl trinitrate cream
- placebo cream (Placebo Comparator): 2 mL of the placebo cream will be placed on the anterior lip of the cervix by a Q-tip applicator, followed by 2 mL will be introduced in the cervical canal 7 minutes prior to IUD insertion
  Interventions: Drug: placebo cream

INTERVENTIONS:
Drug: Lidocaine-Prilocaine cream — 2 mL of the Lidocaine-Prilocaine cream will be placed on the anterior lip of the cervix by a Q-tip applicator, followed by 2 mL will be introduced in the cervical canal 7 minutes prior to IUD insertion
  Arms: Lidocaine-Prilocaine cream
Drug: glyceryl trinitrate cream — 2 mL of the glyceryl trinitrate cream will be placed on the anterior lip of the cervix by a Q-tip applicator, followed by 2 mL will be introduced in the cervical canal 7 minutes prior to IUD insertion
  Arms: glyceryl trinitrate cream
Drug: placebo cream — 2 mL of the placebo cream will be placed on the anterior lip of the cervix by a Q-tip applicator, followed by 2 mL will be introduced in the cervical canal 7 minutes prior to IUD insertion
  Arms: placebo cream

SUMMARY:
the aim of the present study is to compare safety and efficacy of cervical Lidocaine-Prilocaine cream versus glyceryl trinitrate cream on pain perception during levonorgestrel- intrauterine device insertion among nulliparous women: a randomized double-blind controlled trial

ELIGIBILITY:
Inclusion Criteria:

* young and adolescent women requesting LNG-IUD insertion

Exclusion Criteria:

* parous women and contraindications to LNG-IUD placement or to the study drugs.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-10 (Estimated)

PRIMARY OUTCOMES:
pain during LNG-IUD insertion | 5 minutes
  pain during LNG-IUD insertion evaluated by 10 cm Visual analog scale where 0=no pain and 10=worst pain imaginable

SECONDARY OUTCOMES:
duration of the procedure | 10 minutes
  duration of the procedure from speculum in to speculum out